CLINICAL TRIAL: NCT00529919
Title: The Effects of a Weight Loss Diet Containing Medium Chain Triglyceride Oil, Versus Olive Oil, on Body Composition in Free-Living Adults
Brief Title: Effects of Medium Chain Triglyceride Oil, Versus Olive Oil, for Weight Loss
Acronym: Muffin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: International Life Sciences Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F050124003
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Overweight
Keywords: Overweight; Obesity; Weight loss; Medium chain triglycerides; Cardiovascular disease risk
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): MCT oil consumption
  Interventions: Dietary Supplement: Weight loss
- 2 (Placebo Comparator): Olive oil consumption
  Interventions: Dietary Supplement: Weight loss

INTERVENTIONS:
Dietary Supplement: Weight loss — Weight loss study including consumption of either 22-25 g of medium chain triglyceride oil or olive oil
  Other Names: MCT oil, Neobee 1053, Stepan Company

SUMMARY:
The primary aim of this research project is to determine whether the incorporation of food products containing medium chain triglyceride (MCT) oil in a weight-loss program results in a different degree of weight-loss and total and regional fat mass loss than the incorporation of extra light olive oil. The secondary goals are to test whether there are differences in in metabolic risk profile changes between the 2 diets. We hypothesize that men and women who consumed MCT oil as part of their weight loss program will lose more weight and body fat than those who consume olive oil in their weight loss diet.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 27-33 kg/m2
* pre-menopausal women
* weight stable for at least 6 months
* normal score on Brief Symptoms Inventory questionnaire

Exclusion Criteria:

* chronic disease
* weight loss treatment
* medication known to affect body weight
* unstable blood pressure, glucose, lipid levels

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2005-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in body weight and fat mass, change in plasma lipid concentrations, fasting glucose and fasting insulin | 16 weeks

SECONDARY OUTCOMES:
Change in blood pressure, change in fat-free mass | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] St-Onge MP, Bosarge A, Goree LL, Darnell B. Medium chain triglyceride oil consumption as part of a weight loss diet does not lead to an adverse metabolic profile when compared to olive oil. J Am Coll Nutr. 2008 Oct;27(5):547-52. doi: 10.1080/07315724.2008.10719737. PMID 18845704